CLINICAL TRIAL: NCT07289555
Title: Tailored Stapled Single Anastomosis Duodeno-ileal Bypass With Sleeve Gastrectomy (SADI-S): Initial Report and Preliminary Results
Brief Title: Tailored Stapled SADI-S: Initial Report and Preliminary Results
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: El-Sahel Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmed mohamed Yousry, Dr, El-Sahel Teaching Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0307473
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Morbid Obesity; Bariatric Surgery; Malnutrition; Comorbidities
Keywords: SADI-S; Bariatric surgery; Limb length tailoring; Weight loss outcomes; Nutritional status
MeSH Terms: conditions — Obesity, Morbid; Malnutrition | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Single centre, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with morbid obesity (Other): Tailored SADI-S
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Only surgical procedure in the study
  Other Names: SADI-S

SUMMARY:
Obesity is a serious health problem worldwide and can lead to many diseases such as diabetes, high blood pressure, heart disease, and sleep apnea. When lifestyle changes and medications are not enough, metabolic and bariatric surgery (MBS) is currently the most effective and long-lasting treatment option.

This study focuses on one of the newer types of bariatric surgery called Single Anastomosis Duodeno-Ileal Bypass with Sleeve Gastrectomy (SADI-S). This procedure combines two parts:

Sleeve gastrectomy, which reduces the size of the stomach so the patient feels full after eating a small amount.

Duodeno-ileal bypass, which shortens the path food takes through the small intestine to reduce calorie absorption.

Our hospital's surgical team is studying a tailored version of this operation, where the length of the bypassed intestine is adjusted to each patient's anatomy. We believe this personalized approach may improve weight loss results while lowering the risk of vitamin and nutrient deficiencies.

The study will include 40 adult patients with obesity who are undergoing SADI-S surgery, either as their first weight loss operation or as a revision surgery after an earlier sleeve gastrectomy. During the operation, surgeons will measure the total length of each patient's small intestine and use a formula to decide how much of it should be bypassed. The duodeno-ileal connection will be made using a stapled technique, which is expected to be safe and efficient.

After surgery, patients will be followed regularly at 1, 3, 6, 9, and 12 months, and then once per year. At each visit, the study team will monitor weight loss, body mass index (BMI), resolution of diabetes and other obesity-related conditions, nutritional status (including vitamins and minerals), and any side effects such as diarrhea, reflux, or nutritional problems.

The goal of this study is to learn whether this tailored SADI-S technique can provide strong, sustained weight loss and health improvement with fewer long-term complications. The results will help improve surgical planning for future patients by showing whether measuring and customizing the bypass length is safer and more effective than using a fixed length.

All data collected will be kept confidential. Patients' participation in the study will not change their regular care or follow-up, and they can withdraw at any time without affecting their treatment.

DETAILED DESCRIPTION:
Background and Rationale

With obesity rates increasing globally, metabolic and bariatric surgery (MBS) has emerged as the most effective long-term treatment for severe obesity and its related comorbidities such as type 2 diabetes mellitus, hypertension, dyslipidemia, and obstructive sleep apnea. Among the various procedures, laparoscopic sleeve gastrectomy (LSG) and Roux-en-Y gastric bypass (RYGB) have been the most frequently performed worldwide. However, the field continues to evolve with the introduction of newer, simplified techniques that aim to achieve optimal weight loss and metabolic control with lower complication rates and better nutritional safety profiles.

Single-Anastomosis Duodeno-Ileal Bypass with Sleeve Gastrectomy (SADI-S), first described by Sánchez-Pernaute and Torres in 2007, is a simplified derivative of the biliopancreatic diversion with duodenal switch (BPD-DS). This operation combines the restrictive component of sleeve gastrectomy with a single duodenoileal bypass, eliminating one anastomosis compared with the traditional DS. By preserving the pylorus, SADI-S maintains the physiological passage of food and minimizes dumping syndrome, postprandial hypoglycemia, and bile reflux.

Initially, the common channel length was set at 200 cm but was later extended to 250-300 cm to reduce the risk of excessive malabsorption and protein-calorie malnutrition. SADI-S has since demonstrated excellent outcomes in terms of weight loss, diabetes remission, and comorbidity improvement, with acceptable nutritional safety when the bypassed segment is appropriately chosen. The International Federation for the Surgery of Obesity (IFSO) and the American Society for Metabolic and Bariatric Surgery (ASMBS) have both recognized SADI-S as a validated bariatric procedure.

However, despite the growing evidence base, the optimal limb length configuration remains controversial. Most studies use fixed bypass lengths without accounting for wide interindividual variability in total small bowel length (SBL), which can range from 350 to over 1000 cm. Because SBL strongly influences caloric absorption and nutritional outcomes, a "one-size-fits-all" approach may lead to imbalanced results-either inadequate weight loss or excessive malabsorption. Measurement inconsistencies, different starting points for limb calculation, and frequent omission of total SBL assessment further complicate standardization.

Tailoring the bypass limb as a proportion of the measured total bowel length may yield more physiologically balanced results and reduce nutritional complications. Despite concerns that intraoperative measurement prolongs surgery, experienced laparoscopic surgeons can measure SBL efficiently, adding only a few minutes to operative time.

Another point of technical variation in SADI-S relates to the anastomotic technique. The duodeno-ileal anastomosis is technically more demanding than gastrojejunal anastomoses performed in RYGB or OAGB because of the thin duodenal wall and proximity to the pancreas and bile duct. While both hand-sewn and stapled techniques are described, stapled anastomosis is increasingly favored for its reproducibility, shorter operative time, and lower reported rates of leakage and stenosis.

Study Rationale

This prospective observational study aims to evaluate a tailored, stapled SADI-S technique in which the length of the biliopancreatic limb (BPL) is calculated as a fixed percentage (35%) of each patient's measured total small bowel length. By tailoring the limb to each patient's anatomy, the study seeks to optimize outcomes by achieving a balance between sufficient weight loss and nutritional safety.

To our knowledge, this is the first single-center study to systematically assess outcomes using this formula-based approach in stapled SADI-S.

Study Objectives

Primary Objective:

To evaluate the impact of bypassing approximately 35% of the measured total small bowel length on weight loss, nutritional outcomes, and postoperative symptoms in patients undergoing SADI-S (either as a primary or revisional procedure).

Secondary Objectives:

To assess the safety and practicality of using a stapled duodeno-ileal anastomosis in all patients.

To analyze correlations between the tailored BPL length and outcomes such as comorbidity remission, postoperative symptoms, and quality of life.

To assess long-term sustainability of weight loss and rates of nutritional deficiency.

Study Design

This is a prospective, single-center, observational study conducted at the Department of Surgery, El Sahel Teaching Hospital, Cairo, Egypt. The study will include 40 adult patients who meet the inclusion criteria and provide informed consent. Participants will undergo either primary SADI-S or revisional SADI-S after previous sleeve gastrectomy, depending on individual indication.

All surgeries will be performed by experienced bariatric surgeons using a standardized five-port laparoscopic approach.

Preoperative Assessment

All candidates will undergo thorough preoperative evaluation, including:

Complete medical history and physical examination.

Anthropometric measurements: height, weight, BMI.

Laboratory testing: fasting glucose, HbA1c (for diabetics), CBC, liver and renal function tests, coagulation profile, thyroid function, and micronutrient baseline panel.

Cardiopulmonary assessment with ECG and echocardiography.

Upper abdominal ultrasound to detect gallstones; concomitant cholecystectomy will be performed when indicated.

For revisional cases, CT virtual gastroscopy and gastric volumetry to assess sleeve anatomy, pouch volume, and exclude twist or stenosis.

Surgical Technique

1. Patient Positioning and Setup The operation will be performed laparoscopically using a standard five-port configuration. The patient is positioned in the French (split-leg) position with reverse Trendelenburg tilt.
2. Sleeve Gastrectomy Component

   In primary cases, a 50 French bougie is used for calibration, with complete fundus mobilization and linear stapling from the antrum to the angle of His.

   In revisional cases, complete adhesiolysis and pouch resizing are performed, again calibrated over a 50 French bougie.
3. Intraoperative Measurement of Small Bowel Length

   The total small bowel length (TSBL) is measured from the ligament of Treitz to the ileocecal valve.

   Two atraumatic bowel graspers marked at 5 and 10 cm intervals are used to measure the bowel in fully stretched segments, counting hand-by-hand.

   Markings are placed at 150 cm and 200 cm with clips and sutures to facilitate later localization.

   The measurement is typically completed within 8-10 minutes.
4. Tailoring of Bypass Limb

   The biliopancreatic limb (BPL) is tailored to equal approximately 35% of the TSBL.

   For patients with TSBL ≤ 480 cm, a fixed 300 cm common limb is retained to avoid malnutrition.

   For longer TSBL, the duodeno-ileal anastomosis is created at the point corresponding to 65% of the measured total length from the ileocecal valve.
5. Duodeno-Ileal Anastomosis (Stapled Technique)

   The duodenum is transected 3-4 cm distal to the pylorus using a linear stapler.

   The selected ileal segment is brought in an isoperistaltic orientation.

   A side-to-side, functional end-to-end stapled anastomosis is performed using a 45-mm linear stapler.

   The common enterotomy is closed with a single layer of absorbable running suture.

   Air-leak test is performed routinely.
6. Completion

Hemostasis is confirmed.

Drain placement is selective.

Specimen extraction is performed through the umbilical or left upper port.

Postoperative Management

All patients follow a standardized postoperative pathway:

Early ambulation within 6 hours after surgery.

Liquid diet started on postoperative day 1 and advanced as tolerated.

Discharge typically occurs on postoperative day 2-3.

All patients receive lifelong vitamin and mineral supplementation as per international bariatric guidelines.

Follow-Up Schedule

Patients are evaluated at:

1, 3, 6, 9, and 12 months postoperatively, then annually.

At each follow-up, data collected include:

Weight, BMI, and percent excess weight loss (%EWL).

Comorbidity evaluation (diabetes, hypertension, dyslipidemia, sleep apnea, PCOS).

Nutritional laboratory profile (Hb, albumin, vitamin D, calcium, phosphorus, magnesium, ferritin, vitamin B12).

Assessment of gastrointestinal symptoms (reflux, diarrhea, flatulence, dumping, bile reflux).

Quality of life assessment and dietary adherence.

Outcome Measures

Primary Outcomes:

Weight loss effectiveness at 6 months, 1 year, and annually thereafter.

Incidence of postoperative gastrointestinal symptoms.

Secondary Outcomes:

Nutritional outcomes and their correlation with bypassed bowel length.

Resolution rates of metabolic comorbidities.

Safety and feasibility of the stapled duodeno-ileal anastomosis technique.

Data Collection and Analysis

All data will be recorded in a prospective electronic database. Weight loss metrics will be analyzed using %EWL and %TWL. Nutritional markers will be compared across time points and correlated with limb length ratios. Complications will be classified according to the Clavien-Dindo scale.

Continuous variables will be expressed as mean ± SD and analyzed using paired or unpaired t-tests as appropriate. Categorical variables will be analyzed using chi-square tests. Statistical significance will be set at p < 0.05.

Potential Risks and Benefits

The surgical risks are consistent with standard laparoscopic bariatric procedures and include bleeding, leakage, infection, bowel obstruction, and nutritional deficiencies. However, tailoring the bypass length to individual bowel anatomy is expected to lower the risk of severe malabsorption while maintaining adequate weight loss.

Patients are expected to benefit from improved obesity-related comorbidities, enhanced quality of life, and a durable weight loss profile.

Confidentiality and Data Sharing

All participant data will be de-identified and stored securely. Only authorized investigators will have access to the data.

Individual participant data (IPD) will not be shared publicly due to privacy and institutional regulations but may be available upon reasonable request for meta-analyses with ethics approval.

Study Significance

This study represents a step toward personalized bariatric surgery. By objectively measuring bowel length and tailoring the bypass segment, surgeons can minimize variability and optimize outcomes. The use of a stapled anastomosis further standardizes the procedure, reducing technical variability.

If successful, this tailored SADI-S approach could serve as a model for safe, effective, and individualized metabolic surgery, contributing valuable evidence toward standardization of limb length in malabsorptive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* BMI ≥35 kg/m² or BMI ≥30 kg/m² with obesity-related comorbidities such as type 2 diabetes mellitus (T2DM), hypertension, dyslipidemia, obstructive sleep apnea, or non-alcoholic fatty liver disease.
* Willingness to adhere to follow-up visits and testing.
* Indicated for revisional SADI-S post sleeve gastrectomy for inadequate weight loss or weight regain.

Exclusion Criteria:

* Severe uncontrolled medical or psychiatric conditions preventing adherence to the protocol.
* Known short bowel syndrome or previous extensive bowel resections or intraoperative finding of extensive bowel adhesions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss effectiveness | 6 months,1year, 2 years, 3 years, 4 years and 5 years
  Change in weight
Incidence of postoperative symptoms | 6 months,1year, 2 years, 3 years, 4 years and 5 years
  Vomiting, diarrhea, weakness, etc.

SECONDARY OUTCOMES:
Nutritional status and its correlation with limb length | 6 months,1year, 2 years, 3 years, 4 years and 5 years
  Albumin, Na, K, vitamens, etc.
Safety of stapled anastomosis | 6 months,1year, 2 years, 3 years, 4 years and 5 years
  Anastomosis related complications will include postoperative bleeding requiring intervention (via vital signs, CBC, or imaging), confirmed anastomotic or staple-line leakage or anastomotic stenosis (via imaging or endoscopy) requiring endoscopic or surgical treatment. Results will be reported as the number and percentage of participants who experience ≥1 complication.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Yousry, Lecturer of Surgery, Principal Investigator — El Sahel Teaching Hospital, Cairo, Egypt
Locations (1):
- El Sahel Teaching Hospital, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared because this is a single-center observational study with a relatively small sample size (n=40), which may allow indirect identification of participants despite anonymization. However, de-identified summary data and aggregated results supporting the findings of this study will be available from the corresponding author upon reasonable request for academic and non-commercial purposes.

REFERENCES:
- [Background] Man J, Hrabe J. Anastomotic Technique-How to Optimize Success and Minimize Leak Rates. Clin Colon Rectal Surg. 2021 Nov 23;34(6):371-378. doi: 10.1055/s-0041-1735267. eCollection 2021 Nov. PMID 34853557
- [Background] Liagre A, Martini F, Anduze Y, Boudrie H, Van Haverbeke O, Valabrega S, Kassir R, Debs T, Petrucciani N. Efficacy and Drawbacks of Single-Anastomosis Duodeno-Ileal Bypass After Sleeve Gastrectomy in a Tertiary Referral Bariatric Center. Obes Surg. 2021 Jun;31(6):2691-2700. doi: 10.1007/s11695-021-05323-y. Epub 2021 Apr 9. PMID 33834374
- [Background] Salman MA, Abelsalam A, Nashed GA, Yacoub M, Abdalla A. Long Biliopancreatic Limb Roux-En-Y Gastric Bypass Versus One-Anastomosis Gastric Bypass: a Randomized Controlled Study. Obes Surg. 2023 Jul;33(7):1966-1973. doi: 10.1007/s11695-023-06631-1. Epub 2023 May 13. PMID 37178225
- [Background] van der Voort M, Heijnsdijk EA, Gouma DJ. Bowel injury as a complication of laparoscopy. Br J Surg. 2004 Oct;91(10):1253-8. doi: 10.1002/bjs.4716. PMID 15376204
- [Background] Mahawar KK, Parmar C, Carr WRJ, Jennings N, Schroeder N, Small PK. Impact of biliopancreatic limb length on severe protein-calorie malnutrition requiring revisional surgery after one anastomosis (mini) gastric bypass. J Minim Access Surg. 2018 Jan-Mar;14(1):37-43. doi: 10.4103/jmas.JMAS_198_16. PMID 28695878
- [Background] Pereira AM, Moura D, Pereira SS, Andrade S, Almeida RF, Nora M, Monteiro MP, Guimaraes M. Beyond Restrictive: Sleeve Gastrectomy to Single Anastomosis Duodeno-Ileal Bypass with Sleeve Gastrectomy as a Spectrum of One Single Procedure. Obes Facts. 2024;17(4):364-371. doi: 10.1159/000539104. Epub 2024 May 27. PMID 38801818
- [Background] Brown WA, de Leon Ballesteros GP, Ooi G, Higa K, Himpens J, Torres A, Shikora S, Kow L, Herrera MF; IFSO appointed task force reviewing the literature on SADI-S/OADS. Single Anastomosis Duodenal-Ileal Bypass with Sleeve Gastrectomy/One Anastomosis Duodenal Switch (SADI-S/OADS) IFSO Position Statement-Update 2020. Obes Surg. 2021 Jan;31(1):3-25. doi: 10.1007/s11695-020-05134-7. Epub 2021 Jan 6. PMID 33409979
- [Background] Gazer B, Rosin D, Bar-Zakai B, Willenz U, Doron O, Gutman M, Nevler A. Accuracy and inter-operator variability of small bowel length measurement at laparoscopy. Surg Endosc. 2017 Nov;31(11):4697-4704. doi: 10.1007/s00464-017-5538-5. Epub 2017 Apr 13. PMID 28409379
- [Background] Madan AK, Harper JL, Tichansky DS. Techniques of laparoscopic gastric bypass: on-line survey of American Society for Bariatric Surgery practicing surgeons. Surg Obes Relat Dis. 2008 Mar-Apr;4(2):166-72; discussion 172-3. doi: 10.1016/j.soard.2007.08.006. Epub 2007 Dec 19. PMID 18069071
- [Background] Tacchino RM. Bowel length: measurement, predictors, and impact on bariatric and metabolic surgery. Surg Obes Relat Dis. 2015 Mar-Apr;11(2):328-34. doi: 10.1016/j.soard.2014.09.016. Epub 2014 Sep 30. PMID 25614357
- [Background] Kallies K, Rogers AM; American Society for Metabolic and Bariatric Surgery Clinical Issues Committee. American Society for Metabolic and Bariatric Surgery updated statement on single-anastomosis duodenal switch. Surg Obes Relat Dis. 2020 Jul;16(7):825-830. doi: 10.1016/j.soard.2020.03.020. Epub 2020 Mar 30. No abstract available. PMID 32371036
- [Background] Ferraris RP. Dietary and developmental regulation of intestinal sugar transport. Biochem J. 2001 Dec 1;360(Pt 2):265-76. doi: 10.1042/0264-6021:3600265. PMID 11716754
- [Background] Sanchez-Pernaute A, Herrera MA, Perez-Aguirre ME, Talavera P, Cabrerizo L, Matia P, Diez-Valladares L, Barabash A, Martin-Antona E, Garcia-Botella A, Garcia-Almenta EM, Torres A. Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S). One to three-year follow-up. Obes Surg. 2010 Dec;20(12):1720-6. doi: 10.1007/s11695-010-0247-3. PMID 20798995
- [Background] Clapp B, Ponce J, Corbett J, Ghanem OM, Kurian M, Rogers AM, Peterson RM, LaMasters T, English WJ. American Society for Metabolic and Bariatric Surgery 2022 estimate of metabolic and bariatric procedures performed in the United States. Surg Obes Relat Dis. 2024 May;20(5):425-431. doi: 10.1016/j.soard.2024.01.012. Epub 2024 Feb 1. PMID 38448343
- [Background] Eisenberg D, Shikora SA, Aarts E, Aminian A, Angrisani L, Cohen RV, de Luca M, Faria SL, Goodpaster KPS, Haddad A, Himpens JM, Kow L, Kurian M, Loi K, Mahawar K, Nimeri A, O'Kane M, Papasavas PK, Ponce J, Pratt JSA, Rogers AM, Steele KE, Suter M, Kothari SN. 2022 American Society of Metabolic and Bariatric Surgery (ASMBS) and International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) Indications for Metabolic and Bariatric Surgery. Obes Surg. 2023 Jan;33(1):3-14. doi: 10.1007/s11695-022-06332-1. PMID 36336720